CLINICAL TRIAL: NCT03430427
Title: Brain Networks and Mobility Function: B-NET
Acronym: B-NET
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00046460; 1R01AG052419-01A1 (NIH)
Record Dates: First submitted 2018-01-26; First posted 2018-02-12 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Central Nervous System; White Matter Disease
Keywords: BNET; Brain Networks; Mobility Function; SMCCS
MeSH Terms: conditions — Leukoencephalopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, and DNA will be retained for later analysis and for future research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Community-Dwelling Older Adults: The group will consist of 240 community-dwelling older adults with a range of mobility function based on the short physical performance battery (SPPB).

SUMMARY:
Rapidly accumulating evidence indicates that the central nervous system (CNS) plays a pivotal role in mobility function with age-associated CNS changes strongly contributing to declining mobility. Studies linking the brain to mobility have used anatomical measures like brain volume and white matter integrity, and suggest that damage to the connecting fibers of the brain (white matter) is related to mobility impairment. Unfortunately, age-related structural white matter damage appears irreversible and only indirectly indicates the functional connectivity between brain regions. It is believed that functional brain network analyses have the potential to identify individuals that may benefit from interventions prior to the development of irreversible white matter lesions. The current project will assess both physical and cognitive function and integrate these variables with measures of brain network connectivity.

DETAILED DESCRIPTION:
Studies linking the brain to mobility have used anatomical measures like brain volume and white matter integrity, and suggest that damage to the connecting fibers of the brain (white matter) is related to mobility impairment. Unfortunately, age-related structural white matter damage appears irreversible and only indirectly indicates the functional connectivity between brain regions. The preliminary data show that directly assessed patterns of functional connectivity correlate with mobility function and can be changed by interventions that improve mobility function. It is not known how changes in CNS functional connectivity relate to changes in mobility, information critical for the design of interventions targeting CNS connectivity to improve mobility impairments. It is clear that structural connectivity underlies functional connectivity, and that structural brain lesions result in altered functional connections. B-NET will assess white matter (WM) disease burden and microstructural changes and relate these changes to functional brain network connectivity. We hypothesize that because sensory motor cortex community structure (SMC-CS) characterizes current brain organization, it will be associated with mobility function independently of anatomical damage markers. Such knowledge may permit earlier identification of persons at high risk for mobility decline and facilitate earlier and better targeted interventions.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling adults aged ≥70 years
* Willing to provide informed consent; ability to communicate with study personnel.

Exclusion Criteria:

* Serious or uncontrolled chronic disease such as:
* Cancer (stage 3 or 4) or having had radiation or chemotherapy in the past year
* Uncontrolled angina
* Heart failure (stage 3-4)
* Respiratory disease requiring the use of oxygen
* Uncontrolled endocrine/metabolic disease (fasting glucose >250mg/dL)
* Liver failure (AST > 40IU/L and/or ALT > 44 IU/L)
* Renal failure requiring dialysis
* Clinically diagnosed neurologic diseases: Parkinson's disease; Amyotrophic Lateral Sclerosis (ALS); Multiple Sclerosis, prior stroke with residual effects lasting longer than 24hrs
* Diagnosis of schizophrenia, bipolar, or other psychotic disorder
* Diagnosis of Alzheimer's disease or evidence of impaired cognitive function
* Prior traumatic brain injury with residual deficits
* Unwilling or unable to have an MRI brain scan (see MRI screening form).
* Dependent on a walker or another person to ambulate.
* Plans to relocate in the next 2- 3 years.
* Single or double amputee
* Musculoskeletal impairments severe enough to preclude functional testing
* Participating in an exercise or cognitive enhancing intervention
* Any other reason the PI or study physician feels the participant would not adhere to the protocol

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Community-dwelling adults reflecting the gender/race composition of Forsyth County in the target age-range will be identified. The 70 and up age-span was chosen because epidemiologic data shows accelerating functional decline and increased prevalence of white matter abnormalities across this age-range.
Sampling Method: Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
Change in Extended Short Physical Performance Battery (eSPPB) | baseline and 6, 18, and 30 months
  The expanded Short Physical Performance Battery (eSPPB) is a modified version of a widely used assessment of lower extremity physical function that consists of 3 standing balance tasks held for 10 seconds each (side-by-side, tandem and semi-tandem), two 4-m walk tests to assess usual gait speed, and 5 repeated chair stands. To minimize ceiling effects and maximize overall dispersion of test scores, the eSPPB increases the holding time of the semi- and full-tandem stands to 30 seconds and adds a single leg stand and a narrow walk test of balance (walking at usual pace within lines of tape spaced 20 cm apart). eSPPB scores are continuous and range from 0 to 4, with higher scores indicative of better performance.

SECONDARY OUTCOMES:
Change in Cardiovascular fitness | baseline and 18 and 30 months
  The fast-paced 400M walk protocol will be used.
Change in Digit Symbol Substitution Test (DSST) | baseline and 18 and 30 months
  The WAIS-III Digit Symbol Substitution Test will be used.

OTHER OUTCOMES:
Change in Gait Speed | baseline and 18 and 30 months
  This will be assessed over 4 meters 3 times at usual pace and 3 times at fast pace using an instrumented mat (GAITRite System), which provides data on average step and stride length, initial and terminal double support time, as well as the variability in these measures
Change in lower extremity muscle strength | baseline and 18 and 30 months
  Maximal isokinetic knee extension and flexion strength will be measured using an isokinetic dynamometer
Change in postural sway | baseline and 18 and 30 months
  Postural sway during quiet stance will be assessed from Center-of-Pressure (COP) trajectory data collected at 100 Hz using an Advanced Mechanical Technology Incorporated (AMTI) AccuSway biomechanics force platform.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Kritchevsky, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

REFERENCES:
- See also: Effects of a Motor Imagery Task on Functional Brain Network Community Structure in Older Adults: Data from the Brain Networks and Mobility Function (B-NET) Study — https://pubmed.ncbi.nlm.nih.gov/33477358/
- See also: Corrigendum: Examining the intersection of cognitive and physical function measures: Results from the brain networks and mobility (B-NET) study — https://pubmed.ncbi.nlm.nih.gov/36936506/
- See also: Examining the intersection of cognitive and physical function measures: Results from the brain networks and mobility (B-NET) study — https://pubmed.ncbi.nlm.nih.gov/36819728/
- See also: Associations of physical function and body mass index with functional brain networks in community-dwelling older adults — https://pubmed.ncbi.nlm.nih.gov/37054493/